CLINICAL TRIAL: NCT01480934
Title: A Prospective Evaluation of Posterior Capsule Opacification in Eyes With Diabetes Mellitus -A Case Control Study
Brief Title: Evaluation of Posterior Capsule Opacification in Eyes With Diabetes Mellitus
Acronym: DM & PCO
Status: Completed | Type: Observational
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 01072007
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Development of Posterior Capsule Opacification
Keywords: Diabetes,posterior capsule opacification,case control study
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group:A-cases-Patients with a history of Diabetes Mellitus: (N=75 eyes). The inclusion criteria for group A: Diabetes mellitus was defined as glycosylated haemoglobin (Hb A1c ) levels of 6% or more , use of diabetic medication (oral hypoglycemic agents, insulin injection or diet restriction), or a physician's diagnosis of diabetes.
- Group - B:controls: Patients with uncomplicated age-related cataract who were otherwise healthy constituted the controls(Group:)B (n=75 eyes).

SUMMARY:
To compare the development of posterior capsule opacification (PCO) between eyes with and without a history of diabetes mellitus (DM) after single-piece hydrophobic acrylic intraocular lens (IOL) implantation 4 years postoperatively.Diabetes mellitus would not increase the incidence of PCO at 4 years.

DETAILED DESCRIPTION:
There is a paucity of available literature that prospectively evaluates the development of PCO with the single-piece hydrophobic acrylic IOL implantation in diabetic versus non-diabetic eyes on a long-term basis. Therefore, this study was designed to compare the degree of PCO after cataract surgery between diabetic and age-matched non-diabetic patients. This prospective, observational case control study comprised patients who underwent phacoemulsification .The patients were asked to return for postoperative follow-up visits at 1 month, 1 year and 4 years.

the digital images were analyzed for PCO .

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus was defined as glycosylated haemoglobin (Hb A1c ) levels of 6% or more ,
* use of diabetic medication (oral hypoglycemic agents, insulin injection or diet restriction), or a physician's diagnosis of diabetes.
* Patients with uncomplicated age-related cataract who were otherwise healthy constituted the controls (n=75 eyes).

Exclusion Criteria:

* patients with glaucoma,
* high myopia (axial length > 27.0 mm),
* pseudoexfoliation,
* traumatic cataract,
* subluxated cataract,
* previous ocular surgeries,
* allergy to dilating drops.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who underwent phacoemulsification for age-related cataract
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-06; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Development of Posterior capsule opacification. | 4 years
  This prospective, observational case control study comprised patients who underwent phacoemulsification .Subjects with a history of diabetes mellitus (DM) were designated as cases (n=75 eyes).Inclusion criteria for cases: Diabetes mellitus was defined as glycosylated haemoglobin (Hb A1c ) levels of 6% or more , use of diabetic medication (oral hypoglycemic agents, insulin injection or diet restriction), or a physician's diagnosis of diabetes. Patients with uncomplicated age-related cataract who were otherwise healthy constituted the controls (n=75 eyes).

SECONDARY OUTCOMES:
duration of diabetes, stage of diabetic retinopathy | 4 years
  The stage of diabetic retinopathy and duration of diabetes was correlated with the degree of PCO in the cases group.

CONTACTS AND LOCATIONS:
Overall Officials: Gauri D Shah, M.S, Principal Investigator — Iladevi Cataract &IOL Research Centre